CLINICAL TRIAL: NCT05100927
Title: 3D Free-Breathing Multi-echo Acquisition for Whole-body Water/Fat Separation Utilizing DIXON Method
Brief Title: 3D Free-Breathing Multi-echo Acquisition for Whole-body Water/Fat Separation
Status: Withdrawn | Type: Observational
Why Stopped: PI is leaving the Penn State
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 21-129
Record Dates: First submitted 2021-10-06; First posted 2021-10-29 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteer
Keywords: MRIdian MR-Linac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- An MR pulse sequence developing on the MRIdian system: This a pilot study to assess and optimize an MR pulse sequence that we are developing on the MRIdian system. It is a single-center trial recruiting only normal volunteers. Volunteers may be grouped by anatomic region of assessment.

SUMMARY:
The purpose of this study is to help researchers develop MRI imaging techniques that can provide better information for using MRI to treat cancer. MRI is a non-invasive technique that uses magnetic fields and radio waves to create images of the inside of the body.

The investigators of this study are developing an MRI imaging technique that will help with treatment planning for cancer patients. Specifically, the method investigating will help to calculate how the dose the patient needs to treat his/her/their cancer is distributed. This information is required for prescribing the dose to the patient for their cancer treatment.

DETAILED DESCRIPTION:
Combined magnetic resonance and linear accelerator systems (MR-Linac systems) are a powerful new cancer treatment modality. MR-Linac systems promise improved patient outcomes and decreased side effects compared to conventional radiation therapy (RT) systems. These systems yield exquisite soft tissue imaging, offer imaging during RT delivery, and provide a platform for adaptive RT. However, unlike traditional RT planning with computed tomography (CT) measured in Hounsfield units, the MR signal does not correlate with electron density. Electron density information is required to calculate radiation dose maps for RT planning for adaptive RT.

The MRIdian MR-Linac is a low-field system (0.35 Tesla), which is beneficial for applications in RT because it has less effect on the radiation beam than higher field systems. However, low-field MR systems have imaging challenges compared to high-field MR systems. The resonant frequencies between water and fat at 0.35 Tesla are close and traditional methods of separating these tissues (i.e., DIXON-based methods) are more difficult. Furthermore, spectral-selection of fat is not possible, which means traditional fat saturation methods cannot be used at 0.35T. Currently, neither a fat-saturation sequence nor a multi-echo sequence for fat/water separation is available on the MRIdian MR-Linac system. We propose to implement and test a fat/water separation technique optimized for 0.35T. This sequence will enable sCT generation for MR-only simulation (i.e., RT planning without CT) and adaptive RT.

The original DIXON technique for water/fat separation depends on two signal acquisitions - when the fat and water spins are in-phase and opposed-phase. New DIXON methods are more flexible and enable fat/water separation at echo times that are not directly in- and opposed-phase. At 0.35T, the fat and water spins are slow enough that the first echo (i.e., shortest echo) is a near-in-phase echo. Additional echoes will support a 3-point DIXON reconstruction and B0 mapping for inhomogeneity correction.

The long-term goal of this study is to realize the benefits of MR-guided adaptive RT to decrease toxicity and improve patient outcomes. The specific objective of this study is to develop an MR sequence on the low-field MR-Linac for fat/water separation. For the purposes of Radiation Oncology, multi-echo gradient-echo is a fast method to acquire a 3D stack with a large FOV. The images can be reconstructed using a DIXON-based method to produce multiple image types. The resulting images can be used for sCT, which could greatly assist with auto-contouring methods and adaptive planning on MR-Linac systems. These images are also diagnostically used for functional imaging, specifically Dynamic contrast-enhanced imaging (DCE-MRI), which has shown promise at low field, as well as a non-contrast method magnetic resonance angiography (MRA).

Producing these images requires chemical shift imaging. At low fields, chemical shift imaging is difficult as the spectra of fat and water are very close (52 Hz @ 0.35T as compared to 224 Hz @ 1.5T). Traditional DIXON methods use out-of-phase and in-phase echo times (TEs) to separate fat and water. At 0.35T, these TEs are 9.86ms and 19.7ms, respectively. However, long TEs degrade the signal-to-noise ratio (SNR) and lead to long imaging times, particularly for 3D stacks. In addition, B0 inhomogeneity increases and SNR degrades with longer TEs.

The hypothesis is that at 0.35T, the fat and water spins are slow enough that the first echo (i.e., shortest echo, approximately 1ms) is a near-in-phase echo. Additional echoes will support a 3-point DIXON reconstruction and B0 mapping for inhomogeneity correction. I predict that once this multi-echo gradient echo sequence is implemented on the MRIdian system, it can be used to acquire images that will successfully produce water-only, fat-only, in-phase and opposed-phase images.

ELIGIBILITY:
Inclusion Criteria:

* 1. Any male or non pregnant female age ≥18 but ≤ 100 who is capable of giving informed consent.

Exclusion Criteria:

* 1. A subject will be excluded if he/she/they has/have a contraindication to MR scanning based on screening. Examples of contraindications include:

  1. Aneurysm clip
  2. Implanted neural stimulator
  3. Implanted cardiac pacemaker or auto-defibrillator
  4. Cochlear implant
  5. Ocular foreign body (e.g., metal shavings)
  6. Any implanted device (pumps, infusion devices, etc)
  7. Shrapnel injuries 2. Subjects will be excluded if it is deemed that he/she/they has/have a condition which would preclude use for technical development (e.g. morbid obesity, claustrophobia, etc.) or present unnecessary risks (e.g. pregnancy, surgery of uncertain type, implant etc.).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers from the local community
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-22 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
MR acquisition and reconstruction | 90 minutes
  MR methods will be tested in phantoms and then volunteers. Each volunteer will provide images for up to 5 anatomies. When any anatomy has 3 consecutive imaging sessions that meet qualitative metrics for image quality (absence of artifacts), image contrast (proper weighting MR image) and tissue classification (fat/water separation), approval by the Radiation Oncologist will be sought. The project will be complete when all 5 anatomies have obtained approval.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Traughber, DSc, Principal Investigator — Penn State Cancer Institute

IPD SHARING:
Plan to Share IPD: No